CLINICAL TRIAL: NCT00441415
Title: Efficacy and Safety of Fixed Combination Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel Compared to Clindamycin 0.1% / Benzoyl Peroxide 5% Gel in the Treatment of Acne Vulgaris
Brief Title: Efficacy and Safety of Fixed Combination Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29058
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2008-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

INTERVENTIONS:
Drug: Adapalene BPO

SUMMARY:
The purpose of this study is to demonstrate the non-inferior efficacy of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel when compared to Clindamycin 1% / Benzoyl Peroxide 5% Gel in Subjects with acne vulgaris after a 12-week treatment period.

ELIGIBILITY:
Male or female Subjects of any race, between the age of 12 and 35 years inclusive, with acne vulgaris, meeting specific inclusion/exclusion criteria.

Main inclusion criteria:

1. Male or female Subjects of any race, aged 12 to 35 years inclusive, with facial acne vulgaris,
2. Subjects with a minimum of 20 inflammatory lesions (papules and pustules) on the face,
3. Subjects with a minimum of 30 and a maximum of 100 non-inflammatory lesions (open comedones and closed comedones) on the face, excluding the nose.

Main exclusion criteria:

1. Subjects with acne cystic lesions,
2. Subjects with acne conglobate, acne fulminancy, secondary acne (chloracne, drug-induced acne, etc.).

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 272 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in total lesion count (sum of non inflammatory and inflammatory lesions) at week 12.

SECONDARY OUTCOMES:
Percent change from Baseline in total inflammatory and non inflammatory lesion counts at each intermediate visit
Global severity assessment at each post Baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth ARTHUR, MD — Helendale Dermatology - Rochester NY - 585-266-5420; Alicia BUCKO, MD — Academic Dermatology Associates - Albuquerque NM - 505-247-4220; Paul YAMAUCHI, MD — Clinical Research Specialists, Inc. - Santa Monica CA - 310-828-8887; Steven E. KEMPERS, MD — Minnesota Clinical Study Center - Fridley MN - 763-571-4200; Harald GOLLNICK, MD, Principal Investigator — Otto-von-Guericke University - Magdeburg - Germany; Yvonne FRAMBACH, MD — Universitatsklinikum - Lubeck - Germany; Michael MEURER, MD — Dresden University - Dresden - Germany; Christos ZOUBOULIS, MD — Hautklinik und Immunologisches Zentrum des Städtischen Klinikum - Dessau - Germany; Roland KAUFMANN, MD — Zentrum fur Dermatoligie und Venerologie - Frankfurt - Germany; Thomas SCHWARZ, MD — Klinik fur Dermatologie, Venerologie und Allerologie - Kiel - Germany
Locations (4):
- United States (4):
  - Paul YAMAUCHI, Santa Monica, California
  - Steven E. KEMPERS, Fridley, Minnesota
  - Dr Alicia BUCKO, Albuquerque, New Mexico
  - Elisabeth ARTHUR, Rochester, New York

REFERENCES:
- See also: Related Info — http://www.galderma.com/